CLINICAL TRIAL: NCT00817869
Title: Pilot Cluster Randomised Controlled Trial of Flooring to Reduce Injuries From Falls in Elderly Care Units
Brief Title: The HIP-HOP Flooring Study: Helping Injury Prevention in Hospitalised Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Portsmouth (Other)
Collaborators: The Dunhill Medical Trust (Other); National Osteoporosis Society (Other); University of Sheffield (Other); Health & Safety Laboratory (Other); National Patient Safety Agency (Other Government); Department of Health, United Kingdom (Other Government); Portsmouth Hospitals NHS Trust (Other Government); University of Bath (Other)
Responsible Party: Principal Investigator, Martin Severs, Professor, University of Portsmouth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13247; UKCRN ID: 5735
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Accidental Falls
Keywords: Floors and Floorcoverings; Health Services for the Aged; Fractures, bone; Delirium, Dementia, Amnestic, Cognitive Disorders; Frail Elderly; Aged, 80 and over
MeSH Terms: conditions — Fractures, Bone; Neurocognitive Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- New Flooring (Experimental): Will receive 8.3mm thick floor covering (Omnisports EXCEL) to replace previous floor covering.
  Interventions: Other: New flooring
- Standard Flooring (No Intervention): Ward will remain with standard floor covering. The overlay will have a comparable slip resistance rating to the new flooring. The sub-floor will also be comparable.

INTERVENTIONS:
Other: New flooring — 8.3mm thick vinyl floor covering with foam backing, manufactured by Tarkett and installed by Tyndale Flooring Ltd.
  Other Names: Omnisports EXCEL
  Arms: New Flooring

SUMMARY:
In hospitals, older people can fall and hurt themselves. The investigators want to see if a new type of flooring can help stop people hurting themselves as badly, if they accidentally fall.

DETAILED DESCRIPTION:
We will carry out the study in eight elderly care wards across England. We will first study the wards for up to 6 months. Then, half of the wards will have the new floor laid. Wards will be chosen to receive the new floor, or remain with a standard floor, by chance. The new floor has 'shock-absorbent' properties. We will study all the wards for another 12 months. This will allow us to compare the new flooring with the normal flooring.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to the study area on a participating elderly care ward

Exclusion Criteria:

* none.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
fall-related injury | Study duration = 18 months. Outcome measured for each patient for duration of stay in ward (approx. 30 days).

SECONDARY OUTCOMES:
Number of falls | Study duration = 18 months. Outcome measured for each patient for duration of stay in ward (approx. 30 days).
Unexpected adverse events | Study duration = 18 months. Outcome measured for each patient for duration of stay in ward (approx. 30 days).
Slip resistance of flooring | Measured at 4 time-points over 1.5 years (1 month; 6 months; 12 months; 18 months)
Shock-absorbency of flooring | Measured at 4 time-points over 1.5 years (1 month; 6 months; 12 months; 18 months)
Place of residence (for cost-effectiveness analysis) | Each patient followed-up 3 months post-discharge
Quality of life (for cost-effectiveness analysis) | Each patient followed-up 3 months post-discharge
Number of hospital re-admissions (for cost-effectiveness analysis) | Each patient followed-up 3 months post-discharge
User views (patients and staff) | Collected during 1 year follow-up of intervention sites (months 6 to 18)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Severs, Study Chair — University of Portsmouth; Amy K Drahota, Study Director — University of Portsmouth; Derek Ward, Principal Investigator — University of Portsmouth; Julie Udell, Principal Investigator — University of Portsmouth
Locations (8):
- United Kingdom (8):
  - Ward D1, Queen Alexandra Hospital, Portsmouth, Hampshire
  - Newchurch Ward, St Mary's Hospital, Newport, Isle of Wight
  - Ruby Ward, Ellesmere Port Hospital, Ellesmere Port, Merseyside
  - Ward C5, Diana Princess of Wales Hospital, Grimsby, North East Lincolnshire
  - Granby Ward, Harrogate District Hospital, Harrogate, North Yorkshire
  - Draycott Ward, Weston General Hospital, Weston-super-Mare, Somerset
  - Ward 15, Newcastle Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - Ward 25, York District Hospital, York, Yorkshire

REFERENCES:
- [Background] Drahota A, Gal D, Windsor J, Dixon S, Udell J, Ward D, Soilemezi D, Dean T, Severs M. Pilot cluster randomised controlled trial of flooring to reduce injuries from falls in elderly care units: study protocol. Inj Prev. 2011 Dec;17(6):e7. doi: 10.1136/injuryprev-2011-040154. Epub 2011 Sep 2. PMID 21890580
- [Result] Drahota AK, Ward D, Udell JE, Soilemezi D, Ogollah R, Higgins B, Dean TP, Severs M. Pilot cluster randomised controlled trial of flooring to reduce injuries from falls in wards for older people. Age Ageing. 2013 Sep;42(5):633-40. doi: 10.1093/ageing/aft067. Epub 2013 Jul 17. PMID 23868093
- [Result] Latimer N, Dixon S, Drahota AK, Severs M. Cost--utility analysis of a shock-absorbing floor intervention to prevent injuries from falls in hospital wards for older people. Age Ageing. 2013 Sep;42(5):641-5. doi: 10.1093/ageing/aft076. Epub 2013 Jul 9. PMID 23838763